CLINICAL TRIAL: NCT01287780
Title: Local Gentamicin Application to Reduce Postoperative Infection Rate in Hemiarthroplasty After Fracture of the Proximal Femur: a Randomized Controlled Trial
Brief Title: Local Gentamicin Application to Reduce Postoperative Infection Rate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2010/18054
Record Dates: First submitted 2011-01-25; First posted 2011-02-01 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Surgical Wound Infection
Keywords: Humans; Prostheses and Implants; Gentamicin administration and dosage; Surgical sponges; Treatment outcomes
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Collagen-gentamicin sponges (Active Comparator): Two sponges of collagen-gentamicin will be inserted into the hip immediately before closure of the wound. Each sponge (10 by 10 cm) contains 280 mg of collagen and 130 mg of gentamicin.
  Interventions: Device: Collagen-gentamicin sponge
- No intervention (No Intervention)

INTERVENTIONS:
Device: Collagen-gentamicin sponge — A 10 by 10 cm sponge consisting of 280 mg collagen and 130 mg gentamicin.Two sponges are inserted during hemiarthroplasty surgery, one in the joint and one underneath the fascia at the time of surgical closure.
  Other Names: Gentamicin-collagen sponge; Infection prophylaxis in orthopaedic surgery
  Arms: Collagen-gentamicin sponges

SUMMARY:
The majority of elderly patients with a displaced fracture of the proximal femur are now treated with a hemiarthroplasty. Prosthetic joint infection is a devastating complication, and the infection rate is high in this group of elderly patients. Local application of gentamicin produces high antibiotic concentrations in the wound. The aim of this study is to determine whether locally administered collagen-gentamicin in the joint perioperatively in addition to routine IV prophylaxis with beta-lactam antibiotics can reduce the early postoperative infection rate (< 4 weeks postoperative)after hemiarthroplasty in proximal femoral fractures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of proximal femoral fracture
* Must be planned operated with a prosthesis of the hip

Exclusion Criteria:

* Known allergy to gentamicin
* Ongoing treatment with aminoglycosides
* Reduced renal function
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with postoperatively infection after hemiarthroplasty to evaluate locally administered collagen-gentamicin peroperatively | Within 4 weeks after prosthetic surgery
  A randomized multicentre trial

CONTACTS AND LOCATIONS:
Overall Officials: Finnur Snorrason, Ph.D, Study Director
Locations (5):
- Norway (5):
  - Buskerud Hospital, Drammen, Drammen, Drammen
  - Elverum Hospital, Elverum, Elverum
  - Oslo University Hospital, Ullevål, Oslo, Oslo County
  - Asker and Bærum Hospital, Bærum, Rud
  - Diakonhjemmets Hospital, Oslo

REFERENCES:
- [Derived] Westberg M, Frihagen F, Brun OC, Figved W, Grogaard B, Valland H, Wangen H, Snorrason F. Effectiveness of gentamicin-containing collagen sponges for prevention of surgical site infection after hip arthroplasty: a multicenter randomized trial. Clin Infect Dis. 2015 Jun 15;60(12):1752-9. doi: 10.1093/cid/civ162. Epub 2015 Mar 3. PMID 25737375